CLINICAL TRIAL: NCT04687527
Title: Effect of Vitamin D Levels on Postoperative Pain and Narcotic Analgesia in Patients With Laparoscopic Cholecystectomy
Brief Title: Vitamin D Levels and Postoperative Pain in Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Ökkeş Hakan Miniksar, Assistant Professor, Bozok University
Other Study IDs: 189_2020.03.25_02
Record Dates: First submitted 2020-12-22; First posted 2020-12-29 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Vitamin D Deficiency; Postoperative Pain
Keywords: laparoscopic cholecystectomy; Vitamin D Deficiency; Postoperative Pain
MeSH Terms: conditions — Vitamin D Deficiency; Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The deficiency of vitamin D is common in patients with gastrointestinal system disorders.

Vitamin D has been associated with chronic non-specific musculoskeletal pain and migraines due to anti-inflammatory effects.

This prospective observational study will undergo elective laparoscopic cholecystectomy surgery between 18 and 65 years, is planned to participate in ASA (American Society of Anesthesiologists) 1-3, 90 volunteer patients.

In preoperative evaluation, the remaining 3 ml of blood was centrifuged from the routine received blood to determine the level of vitamin D will be kept.

Postoperative will be applied to patient controlled analgesia to all patients for 24 hours.

To determine the level of postoperative pain, the visual analog scale (VAS) will be used in the clock unit and at the service 6, 12 and 24 hours.

In this study, the investigators aimed to test the hypothesis of relation to pain and opioid consumption in acute postoperative (24 hours) of perioperative low-vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer,
* Between the Ages Of 18-65,
* Least Primary School Graduate,
* Not Using Drugs That May Affect Cognitive Functions,
* Non-Alcohol Substance Use,
* Patients Without Psychiatric and Neurological Disease.

Exclusion Criteria:

* Those with known psychiatric disease and drugs,
* Those with an important cardiovascular or central nervous system disease,
* Patients with pain syndromes or routinely using opioid.

Very urgent patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer patients undergoing elective laparoscopic cholecystectomy surgery by the Department of General Surgery
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
preoperative Vitamin D Level and postoperative pain in patients to undergo laparoscopic cholecystectomy operation | 6 months
  Correlations of preoperative Vitamin D Level between postoperative pain in patients undergoing laparoscopic cholecystectomy.to undergo laparoscopic cholecystectomy operation

SECONDARY OUTCOMES:
preoperative Vitamin D Level and opioid analgesic consumption | 6 months
  Correlations of preoperative Vitamin D Level between opioid analgesic consumption in patients undergoing laparoscopic cholecystectomy.to undergo laparoscopic cholecystectomy operation

CONTACTS AND LOCATIONS:
Overall Officials: Ökkeş Hakan Miniksar, Asist.Prof, Study Chair — YOZGAT BOZOK UNIVERSITY
Locations (1):
- Bozok University Medical Center, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided